CLINICAL TRIAL: NCT01376024
Title: Multicenter Prospective Study on Basal Joint Arthritis of the Thumb
Brief Title: Study on Basal Joint Arthritis Prospective
Acronym: BJAM
Status: Suspended | Type: Observational
Why Stopped: Administrative changes
Sponsor: Columbia University (Other)
Collaborators: Orthopedic Research and Education Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: AAAC0826
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Osteoarthrosis of the Carpometacarpal Joint of the Thumb
Keywords: Carpometacarpal arthritis; Basal joint arthritis; CMC arthritis; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The data in this prospective registry will be used 1) to define which surgical and nonoperative techniques are most effective at providing pain relief, restoring function, are cost effective, and patients are satisfied with their outcomes; and 2) to design focused clinical questions regarding the optimal treatment of basal joint arthritis of the thumb in future randomized controlled trials. There are no interventions or changes in patient care associated with this study.

DETAILED DESCRIPTION:
Basal joint arthritis of the thumb is a common condition associated with considerable morbidity. Many non-operative and operative treatments have been described but few multi-center prospective evidence based trials comparing standard treatments have been done. This continuing search for consensus of best clinical practices has been reviewed in a thorough meta-analysis of operative treatments for basal joint arthritis. Through the systematic collection of data regarding patient-specific characteristics, treatment interventions, and longitudinal functional outcome measurements the investigators believe patient outcomes and satisfaction can improve through the elucidation of risk factors for disease progression, and the timing and selection of treatment modalities, either conservative or surgical, for any particular patient. The establishment of a multi-center clinical registry will greatly facilitate these goals.

The study hypothesizes that there exist effective non-operative and operative treatments for certain patient populations with basal joint arthritis of the thumb. There also exists a functionally superior, cost effective, and low risk non-operative or minimally invasive operative treatment regime to alleviate pain and slow the progression of disease in those with less advanced disease. Likewise, there is significant functional, health utility, and economic advantage to surgically treating advanced basal joint arthritis with one of the popularized procedures currently in practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have symptomatic basal joint arthritis.
* Patients who are capable of providing informed consent.

Exclusion Criteria:

* Patients younger than 18 years old at the time of enrollment.
* Patients with neuromuscular disease affecting the operated hand, not caused by the CMC operation.
* Patients with known inflammatory arthritic conditions, such as rheumatoid or psoriatic arthritis.
* Patients with a history of or current infection of the basal joint of the affected hand.
* Patients who are demented or are unable to provide informed consent.
* Patients unable to comply with study guidelines.
* Patients who have metacarpophalangeal joint hyperextension are NOT excluded. These patients will be followed and if they receive a capsulodesis or other procedure at the MCPJ at the same time as their basal joint arthroplasty this will be noted in their data records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study subject population will consist of patients who are diagnosed with CMC arthritis of the thumb stages I, II, III, or IV. Recruitment of subjects will be the responsibility of the operating surgeon or a member of his clincal staff.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2007-03-02 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Flexion/extension range of MCP joint | Baseline, 6 weeks, 3 months, 6 months, 1 year
  Range of motion measured in degrees of the metacarpophalangeal (MCP) joint.
Flexion/extension range of IP joint | Baseline, 6 weeks, 3 months, 6 months, 1 year
  Range of motion measured in degrees of the interphalangeal (IP) joint.
Grip strength | Baseline, 6 weeks, 3 months, 6 months, 1 year
  This will be quantified with use of a Jamar dynamometer set in the second position.
Key-pinch strength | Baseline, 6 weeks, 3 months, 6 months, 1 year
  A 30-lb pinch dynamometer will used to determine lateral key-pinch strength.
Tip-pinch strength | Baseline, 6 weeks, 3 months, 6 months, 1 year
  A 30-lb pinch dynamometer will used to determine lateral tip-pinch strength.

SECONDARY OUTCOMES:
Average total costs per patient | Up to 1 year
  Review or estimation of hospital and office bills including those for the prescribed therapy and/or splinting will be tallied for each patient.
Disability of Arm, Shoulder and Hand (DASH) score | Baseline, 6 weeks, 3 months, 6 months, 1 year
  A questionnaire designed to assess musculoskeletal disorders of the upper limbs.
SF-36 questionnaire score | Baseline, 6 weeks, 3 months, 6 months, 1 year
  A questionnaire designed to validate general health: surveys physical functioning, performance in a physical role, performance in an emotional role, vitality, social functioning, bodily pain, general health perceptions, and mental health.
Prevalence of arthritis progression | Baseline, 6 weeks, 3 months, 6 months, 1 year
  Radiographs will be performed classify each patient within the Eaton 102 osteoarthritis staging system. Sequential radiographs will be examined for progression of joint abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Melvin P Rosenwasser, MD, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University/NY Presbyterian Hospital, New York, New York
  - Vanderbilt University Hospital, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martou G, Veltri K, Thoma A. Surgical treatment of osteoarthritis of the carpometacarpal joint of the thumb: a systematic review. Plast Reconstr Surg. 2004 Aug;114(2):421-32. doi: 10.1097/01.prs.0000131989.86319.b1. PMID 15277809